CLINICAL TRIAL: NCT00202722
Title: Remifentanil as Analgesia for Labour Pain
Brief Title: Remifentanil as Intravenous Patient-controlled Analgesia (IVPCA) During Labour
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSHF812310
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-05

CONDITIONS: Labour Pain; Satisfaction; Adverse Effects
Keywords: Remifentanil, parenteral opioids, obstetric analgesia, IVPCA
MeSH Terms: conditions — Labor Pain; Personal Satisfaction | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Remifentanil IVPCA (Active Comparator): Bolus dose steps of 0.15 microgr/kg, with a 2-min lock-out time
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Intravenous patient controlled analgesia (ivpca) during labour
  Other Names: Ultiva

SUMMARY:
Remifentanil is a ultra short-acting synthetic opioid. It is rapidly metabolized by non-specific blood and tissue esterases. We wanted to investigate the efficacy and safety of remifentanil used as analgesia during labour. Intravenous patient controlled analgesia (ivpca) were used to administer remifentanil. Doses used were 0,15-1,05 mikrogr/kg, with a lock-out time of 2 minutes. 41 women were included in the study. Blood-pressure, heartrate, SaO2, respiration rate and sedation were recorded every 15.minute. Fetal heart rate was recorded for the whole periode of treatment (CTG, STAN). Vaginal contraction pain were assessed by the parturients every 15.minute using a Visual Analogue Scale (VAS). Midwives also recorded their impression of the parturients pain. The parturients level of sedation were recorded by anesthesiologist and midwife every 15.minute. Apgar scores were registered at 1, 5 and 10 min after delivery. Umbilical cord blood analysis regarding blood gases and concentration of remifentanil were performed. After delivery, both mother and midwife evaluated efficacy and safety; Global satisfaction score, if the remifentanil doses were sufficient, nausea, vomiting, level of sedation and dizziness.

DETAILED DESCRIPTION:
Primary and secondary outcome measures presented under "results"

ELIGIBILITY:
Inclusion Criteria:

Healthy women (ASA I-II), in active labour, one fetus with no suspected pathology, expecting normal childbirth, informed consent.

Exclusion Criteria:

Failure to obtain informed consent, received opioids within last 8 hours before study start, serious side-effects mother and abnormal fetal heart rate.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-01; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan H. Rosland, Professor, Study Chair — part time
Locations (1):
- Sorlandet sykehus HF, Kristiansand, Vest-Agder, Norway

REFERENCES:
- [Background] Blair JM, Hill DA, Fee JP. Patient-controlled analgesia for labour using remifentanil: a feasibility study. Br J Anaesth. 2001 Sep;87(3):415-20. doi: 10.1093/bja/87.3.415. PMID 11517125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at arrival to the Labour department
Groups:
- Effect and Side Effects of Remifentanil: Analgesic efficacy and side offects of remifentanil during labour and delivery
Period: Overall Study
Arm/Group | Effect and Side Effects of Remifentanil
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Women in Labour Given Remifentanil Analgesia: Administration of remifentanil analgesia startet with cervical dilatation > 4 cm
Arm/Group | Women in Labour Given Remifentanil Analgesia
Number analyzed (Participants) | 41
Age, Continuous [Mean (Full Range); unit: years] | 27 [20 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Region of Enrollment [Number; unit: participants]
  Norway | 41

OUTCOME MEASURES:

1. Primary Outcome: Pain Score, Visual Analogue Scale (VAS) (Mean Maximal Change in Pain)
Description: Continuous Visual Analogue Scale 0 - 100 millimeters (0=no pain, 100=worst imaginable pain) Registration of pain scores before start and every 15.minute during treatment with remifentanil. Result given is the maximal change in pain score (mean) compared to the baseline value at the given timepoints.
Time Frame: From start with remifentanil treatment until delivery, up to 8 hours.
Population: Per protocol
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Remifentanil: Pain scores
  Satisfaction
Arm/Group | Remifentanil
Number analyzed (Participants) | 41
millimeters | 47 (20.2) [60 to 93]

2. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with remifentanil pain relief by use of questionnaire answered within 24 hours after delivery. Evalutated by a 5-point scale; 1-very satisfied.......5-very dissatisfied.
Time Frame: From start of remifentanil treatment until delivery
Measure: Number; unit: Participants
Groups:
- Satisfaction With Remifentanil Analgesia: Patient satisfaction with remifentanil pain relief by use of questionnaire (within 24-hours after delivery)
Arm/Group | Satisfaction With Remifentanil Analgesia
Number analyzed (Participants) | 41
Participants | 37

ADVERSE EVENTS:
Time Frame: From start of remifentanil analgesia until delivery
Description: Continuous monitoring of oxygen saturation
Groups:
- Maternal Oxygen Desaturation: Oxygen saturation lower than 92% during labour and delivery
Arm/Group | Maternal Oxygen Desaturation
Serious Adverse Events (participants affected / at risk) | 11/41
Other Adverse Events (participants affected / at risk) | 22/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Oxygen Desaturation (N=41)
Oxygen saturation lower than 92% (Respiratory, thoracic and mediastinal disorders) | 11 (11) — Oxygen saturation lower than 92% during labour and delivery, administration of supplemental oxygen
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Oxygen Desaturation (N=41)
Maternal sedation (Nervous system disorders) | 22 (22) — The participants evaluation of sedation level during remifentanil treatment by use of questionnaire within 24 hours after delivery (1=no sedation, 5=very sedated).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No